CLINICAL TRIAL: NCT00854256
Title: Comparison of Canaloplasty and Trabeculectomy in Patients With Open Angle Glaucoma and Inadequate Local Eye Pressure Lowering Therapy - a Prospective, Randomized Study
Brief Title: Trabeculectomy Versus Canaloplasty to Treat Glaucoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Cologne (Other)
Collaborators: iScience Interventional Corporation (Industry)
Responsible Party: Gerhard Welsandt, MD, University of Cologne
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: iScience-022-CG
Record Dates: First submitted 2009-03-02; First posted 2009-03-03 (Estimated); Last update posted 2013-04-15 (Estimated); Status verified 2013-04

CONDITIONS: Glaucoma
Keywords: glaucoma
MeSH Terms: conditions — Glaucoma | interventions — Trabeculectomy; Mitomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Canaloplasty (Experimental)
  Interventions: Procedure: Canaloplasty
- Trabeculectomy with mitomycin C (Active Comparator)
  Interventions: Procedure: Trabeculectomy with mitomycin C

INTERVENTIONS:
Procedure: Canaloplasty — Canaloplasty surgery
  Arms: Canaloplasty
Procedure: Trabeculectomy with mitomycin C — Trabeculectomy with mitomycin C surgery
  Arms: Trabeculectomy with mitomycin C

SUMMARY:
The aim of the study is to investigate pressure lowering effect of two surgical methods canaloplasty and trabeculectomy in patients with open angle glaucoma, in which under local pressure lowering therapy the progression of the disease could not be stopped, and thus a pressure lowering surgical intervention is necessary. The risks in the postoperative course in Canaloplasty in the literature as lower than for the trabeculectomy with mitomycin-C. Conversely, large glaucoma centers questioning the effectiveness of permanent pressure lowering of canaloplasty. Precisely this question is investigated in the study.

ELIGIBILITY:
Inclusion Criteria:

* patients with open angle glaucoma and excavation of 0.4 - 0.8
* 60 eyes of 60 patients (30 patients for trabeculectomy, 30 patients for Canaloplasty) The ratio of female / male is not involved.
* Eye pressure under local therapy: 20mmHg and above (corrected with pachymetry table).
* Local drug therapy: at least 2 eye pressure lowering ingredients or absolute intolerance to preservatives or eye drops.
* general anesthesia possible.
* The operation must be signed by the surgeon as a state-of-the-art performed without complication to be evaluated. If the operation does not meet this criterion, the patient is excluded from the study.

Exclusion Criteria:

* all patients are not included in the group of inclusion criteria, or:
* Phenprocoumon therapy.
* operation is not done state-of-the-art.
* after the surgery: additional eye pressure lowering surgery, cataract surgery, keratoplasty, laser surgery in the anterior eye segment (except suture lysis after trabeculectomy)
* Uveitis, or possible inflammation of the eye
* Previous eye pressure lowering operations or laser interventions
* Corneal Refractive Surgery (pseudophakia allowed)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2009-04; Primary Completion 2013-12 (Estimated); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
Eye pressure | Within 12 month after surgery
  Eye pressure is measured after 1 month, 2 months, 3 months, 6 months, 9 months, and 12 months after surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre of Ophthalmology, University of Cologne, Cologne, North Rhine-Westphalia, Germany